CLINICAL TRIAL: NCT02642809
Title: A Pilot Study Combining Pembrolizumab With Locally Delivered Radiation Therapy for the Treatment of Metastatic Esophageal Cancers
Brief Title: Pembrolizumab With Locally Delivered Radiation Therapy for the Treatment of Metastatic Esophageal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201603087
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Esophageal Neoplasms; Esophageal Cancer; Cancer of the Esophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — pembrolizumab; Brachytherapy; Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Arm 1: Pembrolizumab and Brachytherapy (Experimental): * Brachytherapy dose=16 Gy delivered in 2 fractions of 8 Gy per fraction, separated by 7-10 days between fractions.
  * Pembrolizumab started within 1 week after completion of brachytherapy administered as an intravenous infusion over 30 minutes. It will be given every 3 weeks.
  * Standard of care endoscopic biopsy will take place at time of enrollment and 2-6 months (optional) after pembrolizumab initiation.
  * Research endoscopic biopsy for 8 consented patients will take place 1-2 weeks after initiation of brachytherapy.
  * Peripheral blood will be collected: Pre-brachytherapy, Post-brachytherapy but pre-pembrolizumab (on day 1), Day 22 after the start of pembrolizumab, 3, 6, and 12 months (+/- 2 weeks) after the start of pembrolizumab, and time of progression
  Interventions: Drug: Pembrolizumab; Radiation: Brachytherapy; Procedure: Endoscopic biopsy; Procedure: Computed tomography-guided biopsy; Procedure: Peripheral blood collection

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: MK-3475; Keytruda
Radiation: Brachytherapy
Procedure: Endoscopic biopsy
Procedure: Computed tomography-guided biopsy
  Other Names: CT-guided biopsy
Procedure: Peripheral blood collection

SUMMARY:
The investigators propose to treat patients with metastatic esophageal cancers and dysphagia with two fractions of brachytherapy followed by pembrolizumab. The brachytherapy is hypofractionated and will provide a radiation dose of sufficient intensity to induce the release of tumor-derived antigens and trigger an antitumor immune response. The simplicity of the design should maximize the chance to examine the hypothesis that radiotherapy can induce an immune response, which can then be augmented by pembrolizumab treatment. Success in this study would provide the impetus to conduct further trials aimed at developing this unique strategy as a more broadly applicable therapeutic option in the treatment of patients suffering from these deadly cancers, and will provide important mechanistic insights into the relationship between radiation treatment and immune therapy augmentation.

Taken together, these data indicate that targeting the PD-1/PD-L1 axis in esophageal cancers in combination with radiation therapy may be a rational treatment strategy for these cancers.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with metastatic esophageal cancer that is deemed a candidate for brachytherapy for local control or treatment of dysphagia as determined by treating physician
* Presence of an evaluable metastatic lesion (locoregional lymph nodes are acceptable)
* At least 18 years of age.
* ECOG performance status 0-2
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 x IULN OR Direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (or ≤ 5 x IULN for patients with liver metastases)
  * Serum creatinine ≤ 1.5 x IULN OR Creatinine clearance by Cockcroft-Gault ≥ 60 mL/min/1.73 m2 for patients with creatinine levels > 1.5 x IULN
  * INR or PT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of a anticoagulants
* Sexually active women of childbearing potential and men must agree to use contraceptive methods prior to study entry, for the duration of study participation, and for 120 days after the last dose of pembrolizumab. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Either enrolled in HRPO# 201107221 ("Tissue and Blood Acquisition for Genomic Analysis and Collection of Health Information for Patients with Gastrointestinal Cancers"), which facilitates the collection of specimens for correlative studies, or consenting to collection of blood and tissue as part of this protocol for research testing.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Received a live vaccine within 30 days prior to the first dose of pembrolizumab. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.
* Currently receiving any other investigational agents, has participated in a study of an investigational agent, or use of an investigational device within 4 weeks of the first dose of pembrolizumab.

Has received systemic therapy within 4 weeks of the first dose of pembrolizumab.

* Known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of MK-3475 and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or other agents used in the study.
* Uncontrolled intercurrent illness that would limit compliance with study requirements. This would include, but is not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, immunosuppression, autoimmune conditions, underlying pulmonary disease, or psychiatric illness/social situations.
* Has an active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 72 hours of study entry.
* Known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected).
* Known history of active TB.
* Known history of HIV (HIV 1/2 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Tolerability of localized esophageal hypofractionated brachytherapy administered in two fractions when combined with pembrolizumab as measured by treatment related adverse events | 30 days after completion of treatment (estimated to be 7 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.

SECONDARY OUTCOMES:
Local antitumor effect of hypofractionated brachytherapy followed by pembrolizumab as determined by endoscopic measurements of change in tumor length | Up to 8 weeks post-pembrolizumab treatment (estimated to be 8 months)
Local antitumor effect of hypofractionated brachytherapy followed by pembrolizumab as determined by esophageal lumen diameter | Up to 8 weeks post-pembrolizumab treatment (estimated to be 8 months)
Local antitumor effect of hypofractionated brachytherapy followed by pembrolizumab as determined by grade of dysphagia per CTCAE criteria. | Up to 8 weeks post-pembrolizumab treatment (estimated to be 8 months)
Systemic efficacy of hypofractionated brachytherapy to the esophagus combined with systemic pembrolizumab on non-radiated metastatic lesions as measured by the total tumor size of all the target lesions as measured by irRC-based criteria | Up to 8 weeks post-pembrolizumab treatment (estimated to be 8 months)
  -At the baseline tumor assessment, the sum of the products of the two largest perpendicular diameters (SPD) of all index lesions (five lesions per organ, up to 10 visceral lesions and five cutaneous index lesions) is calculated. At each subsequent tumor assessment, the SPD of the index lesions and of new, measurable lesions (≥5 x5 mm; up to 5 new lesions per organ: 5 new cutaneous lesions and 10 visceral lesions) are added together to provide the total tumor burden
Progression-free survival (PFS) | Up to 1 year after completion of treatment (estimated to be 12 months)
Overall survival (OS) | Up to 1 year after completion of treatment (estimated to be 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Cliff Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu